CLINICAL TRIAL: NCT00658528
Title: A Randomized Double-Blind Parallel Study of Rabeprazole Extended-Release 50 mg Versus Esomeprazole 40 mg for Healing and Symptomatic Relief of Moderate to Severe Erosive Gastroesophageal Reflux Disease (GERD)
Brief Title: Rabeprazole Extended-Release 50 mg Versus Esomeprazole 40 mg for Healing and Symptomatic Relief of Moderate to Severe Erosive Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-G000-301; 2007-005570-32 (EudraCT Number)
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; erosive GERD; erosive esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Rabeprazole sodium
- 2 (Active Comparator)
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Rabeprazole sodium — Rabeprazole ER 50 mg capsule, taken orally, once daily for 4-8 weeks.
  Other Names: Aciphex
  Arms: 1
Drug: Esomeprazole — Esomeprazole 40 mg capsule, taken orally, once daily for 4-8 weeks.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Rabeprazole extended release (ER) 50 mg versus Esomeprazole 40 mg for healing and symptomatic relief among subjects with erosive gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, parallel-group study. Subjects who meet all the inclusion/exclusion criteria will be randomly assigned to 1 of 2 treatment groups, Rabeprazole ER 50 mg or Esomeprazole 40 mg for the treatment of moderate to severe erosive GERD.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

1. Male or female, ages 18 to 75 years.
2. History of GERD symptoms for at least 3 months immediately before screening.
3. Heartburn for at least 2 days a week for at least 1 month before screening.
4. Esophageal erosions of Los Angeles (LA) grades C or D based on EGD taken within 14 days prior to enrollment.
5. Subjects who are H. pylori negative based on a screening test.
6. Females should be either of non-childbearing potential or of childbearing potential. Females of childbearing potential must have negative pregnancy tests prior to randomization. Female subjects of childbearing potential must agree to use medically acceptable methods of contraception.
7. Subjects must be able to read, write, and understand the language of the symptom diary.

KEY EXCLUSION CRITERIA:

1. Current or a history of esophageal motility disorders.
2. Current or a history of Barrett's esophagus. Current esophageal strictures or esophagitis (known or suspected to be due to etiology other than GERD such as infection or medications).
3. Current or a history of Zollinger-Ellison syndrome and other acid hypersecretory conditions, or current gastric or duodenal ulcer.
4. Current or a history of cancer, with the exception of fully excised skin basal cell carcinoma.
5. Inflammatory bowel disease.
6. Unstable diabetes mellitus.
7. History of esophageal, gastric and duodenal surgery except simple suturing of an ulcer.
8. Subjects who require daily use of nonsteroidal anti-inflammatory drugs (NSAIDs), oral steroids (->;= 20 mg/day prednisone or equivalent), or aspirin (->; 325 mg/day).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1061 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, MD, PhD, Study Director — Eisai Inc.
Locations (71):
- Anaheim, California, United States
- Argentina (7):
  - Isidro Casanova, La Matanza, BUE
  - Ramos Mejía, BUE
  - San Isidro, BUE
  - Capital Federal, CBA
  - Mendoza, MEN
  - Rosario, SFE
  - San Juan, SJN
- Australia (6):
  - Five Dock, New South Wales
  - Carina Heights, Queensland
  - Kippa-Ring, Queensland
  - Box Hill, Victoria
  - Frankston, Victoria
  - Malvern, Victoria
- Bulgaria (4):
  - Plovdiv, Bulgaria
  - Sofia, Bulgaria
  - Stara Zagora, Bulgaria
  - Varna, Bulgaria
- Canada (11):
  - Saint John, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Guelph, Ontario
  - Hamilton, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Chile (2):
  - Santiago, Chile
  - Vioa Del Mar, Chile
- Croatia (2):
  - Rijeka, Croatia
  - Zagreb, Croatia
- Tartu, Estonia, Estonia
- France (5):
  - Dieppe, France
  - La Chaussée-Saint-Victor, France
  - Lyon, France
  - Marseille 13, France
  - Nice, France
- Germany (10):
  - Mannheim, Baden-Wurttemberg
  - Munich, Bavaria
  - Hamburg, Hamburg
  - Dietzenbach, Hesse
  - Marburg, Hesse
  - Wiesbaden, Hesse
  - Dortmund, North Rhine-Westphalia
  - Lienen/Kattenve Nne, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Berlin, State of Berlin
- Hungary (9):
  - Budapest, Hungary
  - Dunaújváros, Hungary
  - Kisbér, Hungary
  - Miskolc, Hungary
  - Nagykanizsa, Hungary
  - Nyíregyháza, Hungary
  - Szentes, Hungary
  - Veszprém, Hungary
  - Zalaegerszeg, Hungary
- India (12):
  - Ahmedabad, Gujarat
  - Manipal, Karnataka
  - Bhopal, Madhya Pradesh
  - Aurangabad, Maharashtra
  - Mumbai, Maharashtra
  - Nagpur, Maharashtra
  - Pune, Maharashtra
  - Thane, Maharashtra
  - New Delhi, National Capital Territory of Delhi
  - Ludhiana, Punjab
  - Jaipur, Rajasthan
  - Lucknow, Uttar Pradesh
- Riga, Latvia, Latvia

REFERENCES:
- [Derived] Laine L, Katz PO, Johnson DA, Ibegbu I, Goldstein MJ, Chou C, Rossiter G, Lu Y. Randomised clinical trial: a novel rabeprazole extended release 50 mg formulation vs. esomeprazole 40 mg in healing of moderate-to-severe erosive oesophagitis - the results of two double-blind studies. Aliment Pharmacol Ther. 2011 Jan;33(2):203-12. doi: 10.1111/j.1365-2036.2010.04516.x. Epub 2010 Nov 30. PMID 21114792

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 1061 participants who were randomized, 1055 participants received study treatment.
Groups:
- ESO 40 mg: Esomeprazole (ESO) 40 mg capsule concurrently with placebo (identical in appearance to the RAB Extended Release (ER) 50 mg capsule), once daily for 4 to 8 weeks.
- RAB ER 50 mg: Rabeprazole (RAB) Extended Release (ER) 50 mg capsule concurrently with placebo (identical in appearance to the ESO 40 mg capsule), once daily for 4 to 8 weeks.
Period: Overall Study
Arm/Group | ESO 40 mg | RAB ER 50 mg
Started | 531 (Treated) | 524 (Treated)
Completed | 491 | 479
Not Completed | 40 | 45
Not completed — Adverse Event | 5 | 7
Not completed — Lost to Follow-up | 14 | 22
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Withdrawal of consent | 5 | 6
Not completed — Other | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- ESO 40 mg: ESO 40 mg capsule concurrently with placebo (identical in appearance to the RAB ER 50 mg capsule), once daily for 4 to 8 weeks.
- RAB ER 50 mg: RAB ER 50 mg capsule concurrently with placebo (identical in appearance to the ESO 40 mg capsule), once daily for 4 to 8 weeks.
- Total: Total of all reporting groups
Arm/Group | ESO 40 mg | RAB ER 50 mg | Total
Number analyzed (Participants) | 531 | 524 | 1055
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (13.09) | 48 (13.38) | 48.5 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 202 | 408
  Male | 325 | 322 | 647

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Who Achieved Diary-recorded Sustained Resolution of Heartburn by Week 4
Description: During the first 4 weeks of the Double-blind Phase, participants were to record heartburn in a daily diary. Participant daily symptoms for the assessment of hearburn was based on a commonly used 4-point Likert scale of none, mild, moderate and severe. A participant was considered achieving sustained resolution of heartburn if the participant had maintained at least 7 consecutive heartburn-free days.
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | ESO 40 mg | RAB ER 50 mg
Number analyzed (Participants) | 531 | 524
Percentage of Participants
  Yes | 48.2 | 48.3
  No | 46.3 | 44.3
  Missing | 5.5 | 7.4

2. Primary Outcome: Percentage of Participants With Erosive Gastroesophageal Reflux Disease (eGERD) Who Achieved Endoscopically-confirmed Healing by 8 Weeks
Description: Healing at week 4 or 8 were based on improvement of eGERD of the Los Angeles (LA) classification of esophagitis Grade C or D from Baseline. Classifications include:
  Not Present: No breaks (erosions) in the esophageal mucosa (however, edema, erythema, or friability may be present).
  Grade A: One or more mucosal breaks not more than 5 mm in maximum length. Grade B: One or more mucosal breaks more than 5 mm in maximum length, but not continuous between the tops of 2 mucosal folds.
  Grade C: Mucosal breaks continuous between the tops of 2 or more mucosal folds, but involving less than 75% of the esophageal circumference.
  Gread D: Mucosal breaks involving at least 75% of the esophageal circumference.
Time Frame: Baseline and Week 8
Population: Intent-to-Treat (ITT) Population - all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | ESO 40 mg | RAB ER 50 mg
Number analyzed (Participants) | 531 | 524
Percentage of Participants
  Yes | 75 | 80
  No | 20.3 | 14.9
  Missing | 4.7 | 5.2

3. Primary Outcome: Percentage of Participants With eGERD Who Achieved Endoscopically-confirmed Healing by 4 Weeks
Description: Healing at week 4 or 8 were based on improvement of eGERD of the LA classification of esophagitis Grade C or D from Baseline. Classifications include:
  Not Present: No breaks (erosions) in the esophageal mucosa (however, edema, erythema, or friability may be present).
  Grade A: One or more mucosal breaks not more than 5 mm in maximum length. Grade B: One or more mucosal breaks more than 5 mm in maximum length, but not continuous between the tops of 2 mucosal folds.
  Grade C: Mucosal breaks continuous between the tops of 2 or more mucosal folds, but involving less than 75% of the esophageal circumference.
  Grade D: Mucosal breaks involving at least 75% of the esophageal circumference.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | ESO 40 mg | RAB ER 50 mg
Number analyzed (Participants) | 531 | 524
Percentage of Participants
  Yes | 50.3 | 54.8
  No | 47.8 | 42.6
  Missing | 1.9 | 2.7

ADVERSE EVENTS:
Time Frame: For each participant, from the time of administartion of the first dose of study drug up to 30 days after the administration of the last dose of study drug or up to resolution of adverse event or up to approximately 10 weeks.
Description: Data are presented as number of participants with treatment emergent adverse events (serious and non-serious). The analysis was performed using Safety Analysis Set (SAS) defined as all subjects who received at least 1 dose of study drug and had a postbaseline safety assessment.
Arm/Group | ESO 40 mg | RAB ER 50 mg
Serious Adverse Events (participants affected / at risk) | 4/528 | 4/518
Other Adverse Events (participants affected / at risk) | 0/528 | 0/518
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESO 40 mg (N=528) | RAB ER 50 mg (N=518)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No